CLINICAL TRIAL: NCT02353741
Title: Concurrent EGFR-TKIs and Thoracic Radiation Therapy in EGFR Active Mutation for the First Line Treatment of Non-Small Cell Lung Cancer at Stage IV: A Single-arm, Open-label, Single Center, Phase II Trial.
Brief Title: Concurrent EGFR-TKIs and Thoracic Radiation Therapy in Active EGFR Mutation for 1st Line Treatment of Stage IV NSCLC
Acronym: CERTAIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: too slow of recruitmentc
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, The deputy director of oncology department of Xinqiao Hospital, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-001
Record Dates: First submitted 2015-01-16; First posted 2015-02-03 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EGFR-TKIs combined with radiotherapy (Experimental): EGFR-TKIs combined with concurrent thoracic radiotherapy. Receive oral erlotinib 150mg per day with concurrent thoracic radiotherapy, within 2 weeks, pGTV54～60Gy/27～30f/5.5～6w.
  Interventions: Drug: EGFR-TKIs; Radiation: thoracic radiotherapy

INTERVENTIONS:
Drug: EGFR-TKIs — Beginning on day 2 of treatment, receive oral erlotinib 150mg per day.
Radiation: thoracic radiotherapy — From the beginning of EGFR-TKIs, within 2 weeks, receive concurrent thoracic radiotherapy, pGTV54～60Gy/27～30f/5.5～6w.
  Other Names: thoracic radiation

SUMMARY:
This single-arm phase II study aims to study the efficacy of a possible first line treatment that combines epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKIs) with concurrent thoracic radiation therapy for stage IV non-small cell lung cancer (NSCLC) with active EGFR mutation, as well as assessing PFS, OS, tumor response, etc. to verify that this new combinational therapy can benefit short-term and long-term survival of the patients with advanced NSCLC.

DETAILED DESCRIPTION:
Based on NCCN guideline of the epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKIs) such as erlotinib, gefitinib and icotinib as the first line treatment for advanced Non-Small Cell Lung Cancer (NSCLC), the efficacy of EGFR-TKIs in combination with thoracic radiotherapy as the first line treatment for stage IV NSCLC with active EGFR mutation remains unknown. In this single-arm phase II trial, we chose the subjects with stage IV harboring active EGFR mutation,who were treated by EGFR-TKIs combined with radiation therapy. The primary endpoint is 1-year rate of progression-free survival and the second endpoints are overall survival (OS), objective response rate and toxic and side effect. By evaluating them, we expect to find out the evidence that the combination therapy can benefit the short-term and long-term survival of the patients. Meanwhile, via the stratification analysis of tumor biomarker and immune index, we obtain the evidences for the benefits of comprehensive and individual treatment for advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status≤2；
2. Cytologically or pathologically confirmed stage IV NSCLC ( controlled pleural effusion will be eligible) with active EGFR mutation;
3. Estimated survival time more than 3 months;
4. Age older than 18 years and under 75 years;
5. Adequate bone marrow, hepatic, and renal function;AST and ALT≤2.5 times the highest reference value when not associated with hepatic metastases, or ≤5 times when hepatic metastases occur;
6. Without history of therapy for primary and metastatic disease;
7. With pleural effusion but can be controlled;
8. Asymptomatic bone metastases without treatment;
9. Based on fusion images of 4DCT MIP sketch tumors and lymph nodes, and limit the mean lung dose: V20≤25%，V30≤18%，MLD≤14Gy，V5≤60%;
10. M1a or M1b for metastases, and the number of the distant lesions ≤10；
11. Voluntary to participate in this clinical trial and sign the consent form.

Exclusion Criteria:

1. Patients with serious functional damage of important organs;
2. Patients diagnosed adequately with other malignant tumors;
3. Pregnant or lactating women;
4. Patients in an active period of acute or chronic infectious diseases;
5. Patients who are allergic to any drugs or people with allergies;
6. With brain metastases;
7. With bone metastases needing radiotherapy;
8. Patients who participate in other clinical trials concurrently;
9. Uncontrolled pleural effusion which may intervene the radiotherapy to primary tumor in lung;
10. The number of the distant lesions>10；
11. Patients who are considered not eligible for the trial after evaluation by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
1-year rate of progression-free survival | one year after treatment, followed
  1-year rate of progression-free survival

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of study enrollment until the date of death
  Overall survival (OS)
Objective response rate | up to three years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Disease control rate | up to three years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
patients quality of life | up to three years
  Assessed by EORTC-QLQ C30
Failure mode | up to three years
  The number of patients who failed the treatment of EGFR-TKIs with thoracic radiotherapy.
Toxicities associated with combined erlotinib and concurrent thoracic radiotherapy. Assessed by Common Terminology Criteria for Adverse Events(CTCAE) | up to three years
  Assessed by Common Terminology Criteria for Adverse Events(CTCAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China

REFERENCES:
- [Derived] Zheng L, Wang Y, Xu Z, Yang Q, Zhu G, Liao XY, Chen X, Zhu B, Duan Y, Sun J. Concurrent EGFR-TKI and Thoracic Radiotherapy as First-Line Treatment for Stage IV Non-Small Cell Lung Cancer Harboring EGFR Active Mutations. Oncologist. 2019 Aug;24(8):1031-e612. doi: 10.1634/theoncologist.2019-0285. Epub 2019 Apr 30. PMID 31040256